CLINICAL TRIAL: NCT01370980
Title: Collaborative and Seamless Care in Oncology : a Study in Primary Care to Measure and Reinforce Safety and Adherence to Oral Cancer Treatment
Brief Title: Collaborative Seamless Care in Oncology : Measure and Reinforce Safety and Adherence to Oral Cancer Treatment
Status: Completed | Type: Observational
Sponsor: Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Marie Schneider, Dr, Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland
Other Study IDs: 139/10
Record Dates: First submitted 2011-06-03; First posted 2011-06-10 (Estimated); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Cancer
Keywords: Medication Adherence; Patient Compliance; Patient Acceptance of Health Care; Administration, Oral; Cancer; Letrozol; Exemestan; Imatinib; Sunitinib; Nilotinib; Everolimus; Deferasirox
MeSH Terms: conditions — Neoplasms; Medication Adherence; Patient Compliance; Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study population: Adults (18 years old or more) with one of the following oral oncology treatments: letrozole, exémestane, imatinib, sunitinib, nilotinib, evérolimus, déférasirox

SUMMARY:
The purpose of this study is to implement a support interdisciplinary program(oncologists, pharmacists, physicians, nurses, leagues against cancer) of medication adherence to oral oncology treatments. The aim is to ensure continuity of care between professionals,effectiveness of treatment and patient safety.

DETAILED DESCRIPTION:
80 patients will be included in swiss-romande hospitals and private oncologists and followed by thirty study pharmacies. Each refusal and drop-out will be documented. Follow-up duration is 48 weeks, with a motivational interviewing at least every three months. Patient adherence will be assessed electronically by MEMS (Medication Event Monitoring System).

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Treated for a cancer with oral medication (letrozol, exemestan,imatinib, sunitinib, nilotinib, everolimus, deferasirox)
* French speaking

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with cancer treated by oral medication in swiss-romande hospitals and private oncologists, and enrolled in the adherence program in one of the thirty studies pharmacies.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2010-07; Primary Completion 2011-12 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in Medication adherence | 3 months, 6 months, 9 months, 12 months
  MEMS data, completed by informations given in motivational interviewing

SECONDARY OUTCOMES:
Program implementation | 1 year
  Evaluating the implementation of the program in pharmacies
Oncologists, nurses, pharmacists and patients satisfaction | 1 year
  By questionnaire and interviews
Effect of Adverse Drug Reaction (ADR) on medication adherence | 1 year
  By MEMS data and motivational interviewing informations
Change in Adverse Drug Reaction (ADR) | 3 months, 6 months, 9 months, 12 months
  To evaluate the frequency and severity of ADR and the pharmacist's contribution to their management. Data from motivational interviewing.

CONTACTS AND LOCATIONS:
Overall Officials: Bugnon Olivier, Professor, Study Chair — Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland; Lüthi François, Dr, Study Chair — Clinique Bois-Cerf, Lausanne; Schneider Marie-Paule, PhD, Principal Investigator — Policlinique Medicale Universitaire; Chevaux Bernard, Dr, Principal Investigator — Centre Hospitalier Universitaire Vaudois; Troxler Stéphanie, PhD Student, Principal Investigator — Policlinique Medicale Universitaire; Leila Achtari, MD, Principal Investigator — Centre Hospitalier Univeristaire Vaudois
Locations (1):
- Policlinique Médicale Universitaire and Centre pluridisciplinaire d'oncologie, CHUV, Lausanne, Canton of Vaud, Switzerland